CLINICAL TRIAL: NCT04074447
Title: A Real World Study on the Efficacy of Immunodetection Point Inhibitors for Advanced Esophageal Cancer
Brief Title: The Efficacy of Immunodetection Point Inhibitors for Advanced Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, president, Sun Yat-sen University
Other Study IDs: ctDNA-1
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Esophageal cancer is one of the most common malignancies of the digestive system. Esophageal squamous cell carcinoma is the main type of esophageal cancer, accounting for more than 90% of esophageal cancer in China. The 5-year survival rate is about 15%~25%. Many patients with esophageal cancer are initially diagnosed as advanced, and many patients with early initial diagnosis will still relapse and metastasis after radical treatment. Currently, chemotherapy plays a central role in palliative care, but its objective remission rate is only 20-40%, and the median survival is about 8-10 months. However, most of the current phase III studies on targeted drugs for esophageal squamous cell carcinoma have failed, and the treatment of esophageal squamous cell carcinoma has entered the bottleneck stage. Therefore, it is urgent to explore a treatment method that can significantly improve the prognosis of patients with esophageal cancer. In recent years, with the development of biological immunotherapy, immunocheckpoint inhibitors, including pd-1 inhibitors, pd-l1 inhibitors and ctla-4 inhibitors, have achieved significant curative effect and made breakthroughs in the treatment of multiple solid tumors including melanoma, non-small cell lung cancer and kidney cancer. These immunocheckpoint inhibitors have also been tried for esophageal cancer, with initial success in immunotherapy for esophageal cancer. In this observational study, all patients with esophageal cancer who used immunocheckpoint inhibitors in clinical practice were included, without limitation on the number of treatment lines or combinations of different chemotherapy. Through follow-up observation, the purpose of this study was to analyze the efficacy of immunocheckpoint inhibitors for esophageal cancer in the real world, and to explore the differences in the efficacy of immunocheckpoint inhibitors in different stages of treatment, as well as the efficacy of different chemotherapy combinations, so as to provide clinical evidence for the use of immunotherapy for advanced esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant tumors of the digestive system. Esophageal squamous cell carcinoma, or esophageal squamous cell carcinoma for short, is the main type of esophageal cancer, accounting for more than 90% of esophageal cancer in China. The 5-year survival rate is about 15%~25%. Many patients with esophageal cancer are initially diagnosed as advanced, and many patients with early initial diagnosis will still relapse and metastasize after radical treatment. Currently, chemotherapy plays a central role in palliative care, but its objective remission rate is only 20-40%, and the median survival is about 8-10 months. However, most of the current phase III studies on targeted drugs for esophageal squamous cell carcinoma have failed, and the treatment of esophageal squamous cell carcinoma has entered the bottleneck stage. Therefore, it is urgent to explore a treatment method that can significantly improve the prognosis of patients with esophageal cancer.

In recent years, with the development of biological immunotherapy, immunocheckpoint inhibitors, including PD-1 inhibitors, PD-L1 inhibitors and CTLA-4 inhibitors, have achieved significant curative effect and made breakthroughs in the treatment of multiple solid tumors including melanoma, non-small cell lung cancer and kidney cancer. These immunocheckpoint inhibitors have also been tried for esophageal cancer, with initial success in immunotherapy for esophageal cancer. In 2017, Toshihiko Doi et al. reported the research results of esophageal cancer, and screened a total of 83 cases of advanced esophageal cancer or gastroesophageal junction cancer, among which 37 patients had positive PD-L1 expression, with a positive rate of 44.6%. Finally, 23 patients were enrolled, 78% of whom were squamous cell carcinoma, 87% of whom had received second-line or above treatment before, among which more than 90% had received chemotherapy before, and the overall disease response rate was 30%. The overall partial remission rate was 30%, and 28% of the 18 patients with squamous cell carcinoma achieved partial remission . Another from Japan, multicenter single-arm phase Ⅱ clinical trials designed to explore Nivolumab clinical activity in advanced esophageal squamous cell carcinomas. The 65 included patients with esophageal squamous cell carcinoma received at least second-line treatment, but the expression level of pd-l1 was not detected. Sixty-four patients received intravenous Nivolumab, with median OS of 12.1 months, objective remission rate of 17.2% and disease control rate of 42%. However, the jury is still out on whether single immunocheckpoint inhibitors for esophageal cancer should be used in combination with chemotherapy, in the first line or in the back line, or in combination with different chemotherapy regiments.

CtDNA is an endogenous tumor DNA in circulating blood that is free from cells. It is generally believed that ctDNA in the blood of tumor patients mainly comes from the proliferation of tumor cells after necrosis and apoptosis and the release of tumor cells with active proliferation. At present, most studies have proved that there are consistent genetic changes in the DNA of tumor tissue cells and ctDNA. If there are driver gene mutations in the primary or metastatic foci of patients, it is possible to detect the same genetic changes in their plasma free DNA. Therefore, ctDNA is a characteristic tumor biomarker that can be followed qualitatively, quantitatively and dynamically. Immunodetection point inhibitors, including PD-1 inhibitors, PD-L1 inhibitors and CTLA-4 inhibitors, have achieved significant efficacy in a variety of tumors and are expected to change the current treatment status of tumors. However, there is no recognized indicator that can predict the efficacy of immunotherapy for esophageal cancer.

In this observational study, all patients with esophageal cancer who used immunocheckpoint inhibitors in clinical practice were included, without limitation on the number of treatment lines or combinations of different chemotherapy. Through follow-up observation, the purpose of this study was to analyze the efficacy of immunocheckpoint inhibitors for esophageal cancer in the real world, and to explore the differences in the efficacy of immunocheckpoint inhibitors in different stages of treatment, as well as the efficacy of different chemotherapy combinations, so as to provide clinical evidence for the use of immunotherapy for advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age above 18, male or female.
2. patients with esophageal cancer confirmed by pathology through tumor biopsy or puncture tissue.
3. the patient was assessed as untreatable by surgery.
4. patients received second-line or third-line chemotherapy and were treated with immunodetector point inhibitors.
5. the patient had complete preliminary pathological information, tumor site, pathological type and other information.
6. the patient must have adequate tumor tissue or 5-10 FFPE white tablets to provide; After treatment, patients were returned to the hospital for re-examination every 3 treatment cycles, and plasma and peripheral blood samples could be obtained during the whole process.
7. other indicators of the patients met the general clinical trial enrollment conditions.
8. subjects read and fully understand the instructions to patients, and sign the informed consent.

Exclusion Criteria:

1. blood samples cannot be obtained before treatment.
2. the patient has clear infection status.
3. the patient has other serious diseases besides esophageal cancer.

(5) current patients with alcoholism or drug abuse. (6) pregnant female patients. (7) the patient has a clear history of neurological or mental disorders.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 80 patients with advanced esophageal cancer were enrolled. Patients need to be treated with second - or third-line chemotherapy combined with immunocheckpoint inhibitors. 10ml of edta-anticoagulant blood was collected before the first treatment of the enrolled patients, and the blood samples were gently reversed in the anticoagulant tube for several times to fully anticoagulate. The upper plasma and the lower blood cells were centrifuged at 1800g for 10 min within 4 hours, respectively, and stored at -80 ℃ for later use and provide 5-10 tissue white sheets.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of ctDNA content decreased in patients with good therapeutic effect | through study completion, an average of 2 years
  The proportion of patients with good therapeutic effect whose serum ctDNA content decreased (in any follow-up）

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided